CLINICAL TRIAL: NCT02400762
Title: A Prospective Study of the Safety and Efficacy of InQu® Bone Graft Extender in Transforaminal and Posterior Lumbar Interbody Fusion Surgery
Brief Title: Prospective Study of Safety and Efficacy of InQu® Bone Graft Extender in Lumbar Interbody Fusion Surgery
Acronym: Intebody
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ISTO Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ISTO-INQU05-11-14
Record Dates: First submitted 2015-03-16; First posted 2015-03-27 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2016-08

CONDITIONS: Intervertebral Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect on-label safety and efficacy data where InQu Bone Graft Extender is applied to transforaminal lumbar interbody fusion (TLIF) and posterior lumbar interbody fusion (PLIF).

It is expected that this study will contribute to the compilation of clinical data required to demonstrate the ability of InQu to promote safe, effective and timely spine fusion in patients who undergo PLIF or TLIF surgery. The results of this study will lead to further analysis (i.e. comparison to historical data of other marketed bone graft products, as well as, to local bone alone).

DETAILED DESCRIPTION:
The purpose of this study is to collect on-label safety and efficacy data where InQu Bone Graft Extender is applied to transforaminal lumbar interbody fusion (TLIF) and posterior lumbar interbody fusion (PLIF) at multiple clinical sites.

Adverse events, time to fusion and Patient Reported Outcomes(PROs) will be recorded through 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* A subject may be included if s/he meets the following criteria:

  1. ≥18 years of age;
  2. Able to give appropriate informed consent;
  3. Willing and able to meet the proposed follow-up schedule;
  4. Has documented diagnosis of up to, and including, Grade 1 spondylolisthesis and/or degenerative disc disease;
  5. Has given appropriate consent for, and undergoes, standard-of-care transforminal or posterior lumber interbody fusion;
  6. Use of InQu Bone Graft Extender on-label.

Exclusion Criteria:

1. Any prior lumbar fusion surgery;
2. Requires fusion surgery of more than two adjacent levels;
3. Has fusion surgery requiring titanium cages;
4. Has a systemic infection or has infection at the site of surgery;
5. Has a medical condition or requires post-operative medication that, in the opinion of the investigator, may interfere with bony/soft tissue healing;
6. Has any physical, social, psychological or economic condition that, in the opinion of the investigator, may preclude accurate data collection or evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients who have given consent for and who undergo standard-of-care single level transforaminal or posterior lumbar interbody fusion surgery in which InQu Bone Graft Extender is used on-label.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2013-10; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Post-operative bone fusion as measured by lumbar CT scan Bone fusion | 12 months

SECONDARY OUTCOMES:
Adverse Events | Continual post treatment
Need for subsequent surgical intervention at target and/or adjacent level | Continual post treatment

OTHER OUTCOMES:
Oswestry Disability Index v2.0 | Baseline 3, 6, 12 months
Visual Analogue Scale for leg and back pain | Baseline 3, 6, 12 months
Short-Form-36 | Baseline, 12 months
EQ-5D | Baseline 3, 6, 12 months
Post-operative bone fusion as measured by flexion/extension lumbar X-ray. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Michaela H Purcell, Study Director — ISTO Technologies, Inc.
Locations (2):
- United States (2):
  - University of Southern Califirnia, Los Angeles, California
  - William Beaumont Hospital, Royal Oak, Michigan